CLINICAL TRIAL: NCT06860464
Title: Effects of Remote Ischemic Conditioning Combined With Motor Training on Spinal Reflex Modulation in Healthy Young Adults
Brief Title: Remote Ischemic Conditioning and Spinal Reflex Modulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCIRB 23-001021
Record Dates: First submitted 2025-01-23; First posted 2025-03-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy Young Adults
Keywords: Remote ischemic conditioning; Spinal reflex modulation; H-reflex; Balance training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are masked to group assignment (RLIC vs. Sham conditioning)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (RIC) (Experimental): RIC is achieved via blood pressure cuff inflation to at least 20 mmHg above systolic blood pressure to 250 mmHg on the thigh of dominant LE. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 2 - 6.
  Interventions: Behavioral: Remote Ischemic Condtioning (RIC); Behavioral: Balance training
- Sham conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 25 mm Hg on the thigh of the dominant LE. Sham involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. Sham conditioning is performed on visits 2-6.
  Interventions: Behavioral: Sham Conditioning; Behavioral: Balance training

INTERVENTIONS:
Behavioral: Remote Ischemic Condtioning (RIC) — See descriptions under arm/group descriptions. RIC is delivered for 5 intervention visits. Visits 1 is the baseline assessment visit, and visits 2-6 are RIC plus training visits.
  Arms: Remote Ischemic Conditioning (RIC)
Behavioral: Sham Conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 5 intervention visits. Visits 1 is the baseline assessment visit, and visits 2-6 are Sham plus training visits.
  Arms: Sham conditioning
Behavioral: Balance training — All participants will undergo training on a balance board, learning to hold the board level within the 5- degree horizontal range. Participants perform the balance task for 15, 30-second trials per day at visits 2-6.

SUMMARY:
Remote ischemic conditioning (RIC) is a clinically feasible method that protects distant organs from severe injury through brief, sub lethal periods of ischemia followed by re-perfusion. Recent studies suggest that RIC, combined with training, improves muscle strength and balance in healthy adults and post-stroke survivors. While the underlying mechanisms are not fully understood, RIC's neuroprotective effects - such as promoting angiogenesis, neurogenesis, and modulating glutamate and GABA synthesis - overlap with neuroplasticity processes. Evidence indicates that neuroplasticity from exercise training occurs not only in the cerebral cortex but also within the spinal cord, yet the role of spinal reflex mechanisms underlying the benefits of RIC remains under explored. Therefore, this study aims to investigate effects of RIC on spinal reflex modulation in healthy adults, both independently and combined with balance training.

DETAILED DESCRIPTION:
Ischemic conditioning (IC) is an endogenous phenomenon that protects target organs from severe ischemic events by applying alternating cycles of brief, sublethal ischemia followed by reperfusion. Remote ischemic conditioning (RIC) is a more feasible, non-invasive method of delivering IC. It involves using a standard blood pressure cuff on either the arm or leg to induce brief periods of sublethal ischemia. Extensive evidence from both animal and human studies indicates that RIC provides neuroprotection through multifactorial mechanisms involving inflammatory, oxidative, excitotoxic, metabolic, vascular, and glial pathways. Additionally, several studies demonstrate the involvement of peripheral somatosensory, spinal cord, and autonomic pathways in RIC-induced neuroprotection. Prior research also shows that RIC enhances motor learning (balance performance) when paired with motor training in both young and older adults. While a wealth of research has shown that neuroplasticity in response to training occurs in cortical and spinal neural circuits, limited studies have explored the effects of RIC on spinal modulations in healthy adults. Notably, only one study has reported a reduction in Hoffman (H)-reflex amplitudes with RIC. Given the evidence of peripheral neuronal pathways involved in RIC and its positive impact on balance performance, it is plausible that RIC could lead to spinal reflex modulations and enhance balance improvements in healthy adults. These modulations may be further amplified when RIC is combined with balance training. The specific aims of this study are to determine whether 1) remote ischemic conditioning (RIC) combined with balance training modulates spinal reflex excitability, as reflected by H-reflex measures, and 2) to examine whether RIC combined with balance training leads to greater improvements in balance performance compared to sham conditioning combined with training in healthy adults. In this single-blind, randomized controlled trial, 30 healthy adults aged 18-40 years will undergo H-reflex testing of the dominant lower extremity and balance assessments at baseline (pre-training). Participants will then be randomized to receive either RIC or sham conditioning combined with a 5-day balance training program. RIC or sham conditioning will be delivered using cyclic inflation and deflation of a pressure cuff applied to the thigh of the dominant lower extremity following a standardized protocol. Balance training will consist of standing on a stability platform with the goal of maintaining the platform within a 5-degree horizontal range for 30 seconds across 15 trials per day for five consecutive days. All outcome measures, including H-reflex parameters (Hmax, maximal H-reflex amplitude, and Hmax/Mmax ratio) and balance performance, will be reassessed post-training following completion of the 5-day intervention. It is hypothesized that, compared to sham conditioning combined with balance training, RIC combined with balance training will result in greater reductions in H-reflex excitability and greater improvements in balance performance from baseline to post-training. This study will help clarify whether RIC induces alterations in spinal reflex modulations when applied independently or in combination with motor training, thereby reflecting neuroplasticity within the spinal cord in healthy young adults. These findings would deepen our understanding of the spinal mechanisms underlying the benefits of RIC and could accelerate its translation for individuals with neurological disorders

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-40 years of age

Exclusion Criteria:

* Individuals with cognitive deficits or communication problems
* Individuals with impaired vision
* Individuals with balance disorders such as vestibular disorders, etc.
* Individuals who are pregnant
* Individuals with known cardiorespiratory dysfunctions
* Presence of lower extremity condition, injury, or surgery within last three months which could compromise training

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximal H-reflex amplitude (Hmax) | Baseline, Day 7
  The maximal (peak) H-reflex amplitude will be determined from the recruitment (stimulus-response) curve. The Hmax amplitude provides an estimate of the number or proportion of motor neurons (MNs) activated from the total MN pool, reflecting spinal reflex modulations and spinal neuroplasticity.
Change in Hmax/ Mmax Ratio | Baseline, Day 7
  The maximal H-reflex and maximal M-wave amplitudes will be determined from the recruitment curve procedure. Calculating the Hmax/Mmax ratio is a standardization method used to reduce variability in H-reflex amplitude across participants. This provides a better basis for comparison and a more reliable estimate of changes in spinal reflex modulations between participants.

SECONDARY OUTCOMES:
Change in Balance Performance | Baseline, Day 7
  The average amount of time in seconds that a participant maintains the stability platform within ±5° of horizontal position during 15 trials of 30 seconds each. The total score will range between 0-30 seconds. Higher balance score indicates better balance performance. Greater average balance time indicates better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Swati M Surkar, PT, PhD, Principal Investigator — East Carolina University
Locations (1):
- Swati Surkar, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on NIH figshare network and will be made available on request.
Supporting Information: ICF
Time Frame: After publishing the results of the study
Access Criteria: Data will be made available upon request to the principal investigator.

REFERENCES:
- [Background] Taube W, Kullmann N, Leukel C, Kurz O, Amtage F, Gollhofer A. Differential reflex adaptations following sensorimotor and strength training in young elite athletes. Int J Sports Med. 2007 Dec;28(12):999-1005. doi: 10.1055/s-2007-964996. Epub 2007 May 11. PMID 17497570
- [Background] Quadrado IC, Cancio RB, Silva BM, Vianna LC, Mezzarane RA. Modulation of spinal cord excitability following remote limb ischemic preconditioning in healthy young men. Exp Brain Res. 2020 May;238(5):1265-1276. doi: 10.1007/s00221-020-05807-w. Epub 2020 Apr 17. PMID 32303809
- [Background] Surkar SM, Bland MD, Mattlage AE, Chen L, Gidday JM, Lee JM, Hershey T, Lang CE. Effects of remote limb ischemic conditioning on muscle strength in healthy young adults: A randomized controlled trial. PLoS One. 2020 Feb 4;15(2):e0227263. doi: 10.1371/journal.pone.0227263. eCollection 2020. PMID 32017777
- [Background] Dirnagl U, Becker K, Meisel A. Preconditioning and tolerance against cerebral ischaemia: from experimental strategies to clinical use. Lancet Neurol. 2009 Apr;8(4):398-412. doi: 10.1016/S1474-4422(09)70054-7. PMID 19296922
- [Background] Kharbanda RK, Nielsen TT, Redington AN. Translation of remote ischaemic preconditioning into clinical practice. Lancet. 2009 Oct 31;374(9700):1557-65. doi: 10.1016/S0140-6736(09)61421-5. PMID 19880021